CLINICAL TRIAL: NCT03192085
Title: Specificity and Patient Perception of SITA-Standard Compared to SITA-Fast Visual Fields in Patients Suspected of Having Glaucoma
Brief Title: Comparison of SITA-Standard Compared to SITA-Fast Visual Fields.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); University of Plymouth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MS/22/02/17
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Randomised crossover trial of diagnostic test with assessment of comparative accuracy - feasibility study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SITA FAST then SITA STANDARD (Other): SITA FAST and SITA STANDARD
  Interventions: Diagnostic Test: SITA FAST VISUAL FIELD TEST; Diagnostic Test: SITA STANDARD VISUAL FIELD TEST
- SITA STANDARD then SITA FAST (Active Comparator): SITA FAST and SITA STANDARD
  Interventions: Diagnostic Test: SITA FAST VISUAL FIELD TEST; Diagnostic Test: SITA STANDARD VISUAL FIELD TEST

INTERVENTIONS:
Diagnostic Test: SITA FAST VISUAL FIELD TEST — Diagnostic test for glaucoma
Diagnostic Test: SITA STANDARD VISUAL FIELD TEST — Diagnostic test for glaucoma

SUMMARY:
This study will compare SITA-Standard and SITA-Fast tests in patients newly referred to the glaucoma screening clinic at the RD&E hospital.

DETAILED DESCRIPTION:
This study will compare SITA-Standard and SITA-Fast tests in patients newly referred to the glaucoma screening clinic at the RD&E hospital. In addition to standard care (SITA-Fast) each person who agrees to take part in the trial will undertake one extra visual field test (SITA-Standard). By comparing the results of the two types of visual field test the investigators aim to provide information on which of the two tests is more specific for glaucoma and which test is better tolerated by patients. The investigators anticipate that this study will generate sufficient data to support a grant application for a longitudinal study to examine the relative merits of different visual field tests in patients with glaucoma and those suspected of developing the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old attending the West of England Eye Unit Glaucoma Service who have been newly referred for suspected glaucoma.

Exclusion Criteria:

* 1. Patients who are unable to perform visual field tests. 2. Patients who are unable to have a full glaucoma assessment. 3. Patients who have undertaken visual field tests in hospital eye departments in the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
specificity of the visual field tests | 1 year
  specificity

SECONDARY OUTCOMES:
Patients' rating of test difficulty | 1 year
  number
The number of "questions asked" (number of presented stimuli). | 1 year
  number

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smith, MBChB, Principal Investigator — Royal Devon

IPD SHARING:
Plan to Share IPD: No